CLINICAL TRIAL: NCT02630004
Title: Phase IB-II Clinical Trial of Melatonin Oral Gel for the Prevention and Treatment of Oral Mucositis in Patients With Head and Neck Cancer Undergoing Chemoradiation.
Brief Title: Melatonin Oral Gel for Oral Mucositis in Patients With Head and Neck Cancer Undergoing Chemoradiation
Acronym: MUCOMEL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spherium Biomed (Industry)
Collaborators: Institut Català d'Oncologia L'Hospitalet (Unknown); Hospital Universitari de la Vall de Hebron (Unknown); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Institut Català d'Oncologia ICO Girona (Unknown); Institut Català d'Oncologia ICO Badalona (Unknown); Hospital Miguel Servet (Other); Hospital Universitario La Paz (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario Virgen de la Victoria (Other); Hospital San Carlos, Madrid (Other); Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JAN13004-30
Record Dates: First submitted 2015-12-03; First posted 2015-12-15 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Oral Mucositis
Keywords: Mucositis; Head and Neck cancer; Chemoradiation
MeSH Terms: conditions — Stomatitis; Mucositis; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Experimental): Melatonin oral gel 3%
  Interventions: Drug: Melatonin oral gel 3%
- Placebo (Placebo Comparator): Placebo oral gel
  Interventions: Drug: Placebo oral gel

INTERVENTIONS:
Drug: Melatonin oral gel 3%
  Arms: Melatonin
Drug: Placebo oral gel
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the efficacy of melatonin oral gel compared to placebo in the prevention and treatment of oral mucositis in patients with head and neck cancer undergoing concurrent chemoradiation.

Other objectives are to assess the Quality of Life (QoL), to evaluate the safety and tolerability and to assess the pharmacokinetic profile of melatonin oral gel administration, in all cases compared to placebo in patients with head and neck cancer and oral mucositis secondary to concurrent chemoradiation.

DETAILED DESCRIPTION:
The study is designed as a prospective, randomized, double blind and placebo-controlled study.

Eligible patients with head and neck cancer undergoing chemoradiation will be randomized assigned at one-to-one ratio to receive

* Group A: melatonin oral gel 3%
* Group B: placebo

All patients will receive standard symptomatic treatment for oral mucositis along the study according to routine clinical practice of the hospital.

A full PK and safety assessment will be carried out in the first 24 patients included in the study (PK subgroup).

All patients will take melatonin oral gel 3% or placebo oral gel from two to three days before start of systemic treatment until one to four weeks after completion of radiotherapy. In the case of concurrent chemotherapy with cisplatin, patients will remain on study from the first day of chemoradiotherapy during 19 weeks (seven on chemoradiotherapy treatment, a maximum of four weeks after completion of radiotherapy and eight more weeks on observation). In the case of patients receiving cetuximab, since the first infusion of cetuximab will be administered one week before the first day of radiation, the patients will remain on study during 20 weeks (eight weeks on chemoradiotherapy, a maximum of four weeks after completion of radiotherapy and eight more weeks on observation). Investigators should take into account that the minimum duration of the melatonin oral gel 3% treatment would be 8 weeks for patients treated with cisplatin and 9 weeks for patients treated with cetuximab.

Patients with oral mucositis improved to grade 1 (based on RTOG) until one to four weeks after the end of chemoradiation may stop melatonin oral gel 3% or placebo treatments. Patients with grade ≥ 2 oral mucositis at this time-point (four weeks after the end of chemoradiation) will stop treatment per protocol (melatonin or placebo) and will continue with standard treatments and under observation until the last safety visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years or over.
2. Patients who gave written informed consent.
3. Life expectancy ≥ 3 months.
4. Subjects willing to comply with treatment and follow-up.
5. Histologically confirmed diagnosis of non-metastatic TNM-2010 stage III-IV squamous cell carcinoma of the following sites:

   * oral cavity
   * oropharynx
   * or any Head and Neck site with lymph nodes at cervical level II.

   Or histologically confirmed carcinoma of the nasopharynx (differentiated squamous cell carcinoma or NonKeratinizing carcinoma or undifferentiated carcinoma) found eligible for chemoradiation with or without neoadjuvant chemotherapy.
6. Patients who have a treatment plan based on systemic treatment (cisplatin or cetuximab) concurrent with radiation with curative intent. Patients may have received up to 3 cycles of neoadjuvant chemotherapy if local adverse events related to this treatment are fully resolved before study entry. Patients with a plan of postoperative chemoradiation may be included only if the primary tumour is located in the oral cavity.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
8. Adequate baseline organ function (hematologic, liver, renal, nutritional and metabolic):

   * Haematology:

     * Absolute neutrophil count (ANC) ≥1.5 x 109/L
     * Haemoglobin ≥ 10 g/dL
     * Platelets ≥ 100,000 x 109/L
   * Hepatic:

     * Total bilirubin ≤ 2 X (Upper limit normal) ULN
     * Alanine amino transferase (ALT) and Asparatate aminotransferase (AST) ≤5 x ULN
   * Renal:

     * For patients who will receive cisplatin: Serum creatinine ≤ ULN or, if > ULN calculated creatinine clearance (ClCR) ≥ 60 mL/min.
     * For patients who will receive cetuximab: Serum creatinine <2.0 mg/dl.
   * Nutritional and metabolic:

     * Albumin > 3.0 mg/dl
     * Magnesium > lower limit normal (LLN) for patients who will receive cetuximab

Exclusion Criteria:

1. Patients with blistering disease.
2. Patients who require feeding with either nasogastric tube, gastrostomy or jejunostomy at study entry
3. Patients whose radiotherapy treatment planned dose is lower than 66 Gy
4. Patients being receiving another investigational agent because of participation in another therapeutic trial
5. Patients treated with fluvoxamine, estrogens, cimetidine, 5- and 8 methoxypsoralen and/or carbamazepine
6. Active viral, bacterial or fungal infections of the mouth in the last 14 days (i.e. stomatitis related to herpes virus or candida)
7. Pregnancy or lactation
8. Known allergy to melatonin
9. Prior radiotherapy of the head and neck
10. Patients with a treatment plan consisting of chemoradiation followed by further chemotherapy
11. Patients with a diagnostics of a synchronic neoplasia except for non-melanoma skin cancer curable with local treatment or in situ cervix carcinoma
12. Any investigational agent within 30 days prior to inclusion
13. Male or female of childbearing age who do not agree with taking adequate contraceptive precautions, i.e. use contraception double barrier (e.g. diaphragm plus condoms) or abstinence during the course of the study and for 2 months after the last administration of the study drug for women and 1 month for men
14. Psychological, geographical, familial or sociological conditions that potentially prevent compliance with the study protocol and follow-up schedule according to investigator criteria. These conditions should be discussed with the patient before inclusion in the trial.
15. Any other medical condition that would make the patient inappropiate for study participation according to the Investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Number (percentage) of patients who develop severe oral mucositis (grade 3-4 according to the RTOG scale) | up to 19-20 weeks

SECONDARY OUTCOMES:
Number (percentage) of patients who develop severe oral mucositis (grade 3-4 according to NCI-CTCAE) | up to 19-20 weeks
Number of days with mucositis of any grade according to the RTOG scale | up to 19-20 weeks
Number of days with grade 3-4 mucositis according to the RTOG scale | up to 19-20 weeks
Time to onset of grade 3-4 mucositis according to the RTOG scale from starting systemic antineoplastic treatment | up to 19-20 weeks
Change from baseline in EORTC QLQ-C30 and EORTC QLQ-H&N35 scores at 4w after RT start | up to 4-5 weeks
Change from baseline in EORTC QLQ-C30 and EORTC QLQ-H&N35 scores at one week after completion of RT | up to 8-9 weeks
Change from baseline in EORTC QLQ-C30 and EORTC QLQ-H&N35 scores at 3 months after completion of RT or before surgery - if it is required post-chemoradiation due persistent or recurrent disease | up to 19-20 weeks
Change from baseline in ECOG-Performance status score at different time points along the study | up to 19-20 weeks
Number (percentage) of patients with grade 1-4 NCI-CTCAE adverse events related to IMP (melatonin oral gel 3%) | up to 19-20 weeks
Number (percentage) of patients who develop cisplatin or cetuximab-associated grade 1-4 adverse events according to the NCI-CTCAE scale | up to 19-20 weeks
Number (percentage) of patients who develop radiation-associated adverse events different from oral mucositis according to the RTOG scale | up to 19-20 weeks
Pharmacokinetics evaluation [Cmax] | up to 11-12 weeks
Pharmacokinetics evaluation [Tmax] | up to 11-12 weeks
Pharmacokinetics evaluation [AUC] | up to 11-12 weeks
Pharmacokinetics evaluation [T1/2] | up to 11-12 weeks
Pharmacokinetics evaluation [Vd] | up to 11-12 weeks
Pharmacokinetics evaluation [Clearance] | up to 11-12 weeks

OTHER OUTCOMES:
Change from baseline in oral pain intensity measured by VAS at different time points along the study. | two times a week up to 19-20 weeks
Number (percentage) of patients who need minor or major opioids | up to 19-20 weeks
Number (percentage) of patients who need special procedures on nutritional status (feeding tube, jejunostomy, gastrostomy) | up to 19-20 weeks
Radiotherapy treatment breaks (cause) | up to 8-10 weeks
Radiotherapy treatment breaks (number of days) | up to 8-10 weeks
Total dose and intensity of radiotherapy: Total Gy; | up to 8-10 weeks
Total dose and intensity of radiotherapy: Gy/week; | up to 8-10 weeks
Total dose and intensity of radiotherapy: Gy/day | up to 8-10 weeks
Milligrams of systemic antineoplastic treatment administered (dose intensity: mg/m2/week) | up to 8-10 weeks
Number (percentage) of patients with complete response using the RECIST 1.1 criteria | 2 months after completion of radiotherapy
Number (percentage) of patients with partial response using the RECIST 1.1 criteria | 2 months after completion of radiotherapy
Number (percentage) of patients with stable disease using the RECIST 1.1 criteria | 2 months after completion of radiotherapy
Number (percentage) of patients with progression disease using the RECIST 1.1 criteria | 2 months after completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Lozano, MD, Principal Investigator — Institut Català d'Oncologia L'Hospitalet
Locations (11):
- Spain (11):
  - Institut Català d'Oncologia ICO Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de la Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia Girona, Girona
  - Hospital San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided